CLINICAL TRIAL: NCT07200284
Title: Periodontal Air-Polishing Device Reduces Tissue Damage and Improves Clinical Outcomes and Exosomal Modulation. A Randomized Clinical Trial
Brief Title: Periodontal Air-Polishing Device Versus Manual Scaling and Root Planing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marco Bonilla, Research Intern, Dp of Periodontics, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4566/CEIH/2024
Record Dates: First submitted 2025-08-11; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Pulmonary Ventilation

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (manual SRP) (Active Comparator): The gold standard treatment for periodontitis
  Interventions: Procedure: Manual SRP
- Airflow (Experimental): An ultrasonic and air-polishing device for periodontal debridement
  Interventions: Procedure: Airpolishing device

INTERVENTIONS:
Procedure: Airpolishing device — The authors will assess biochemical and clinical variables
  Other Names: Airflow
  Arms: Airflow
Procedure: Manual SRP — Gold standard
  Arms: Control (manual SRP)

SUMMARY:
This study looks at two common ways to perform deep cleaning of the gums in people with periodontitis: Airflow® (a spray system that uses fine powder and water) and hand scaling (cleaning with metal instruments). The investigators want to see how each treatment affects inflammation at the molecular level by measuring exosomes (tiny particles released by cells that carry signals) and cytokines (proteins that help regulate inflammation) in the fluid around the gums.

Participants will receive one of the two standard treatments and will have samples taken from the mouth (saliva and/or gum fluid) at specific times before and after treatment. The authors will also record clinical measurements such as bleeding, gum pocket depth, and attachment loss, as well as simple questionnaires about symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Periodontitis patients

Exclusion Criteria:

* Diabetes or other uncontrolled systemic inflammatory diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-08-11 (Actual)

PRIMARY OUTCOMES:
Bleeding on Probing (BOP) | Pre-treatment and Re-Evaluation (4-6 weeks after treatment)
  Description: Proportion of sites showing bleeding upon gentle probing. Unit of Measure: Percentage (%)
Biochemical variables | Pre-treatment and Re-Evaluation (4-6 weeks after treatment).
  Concentration of exosomes and cytokines using a commercial kit, measured in pg/mL. Gingival Crevicular Fluid will be obtained using the Mombelli technique (introducing an absorbent paper point inside the periodontal pocket)
Periodontal Pocket Depth (PPD) | Pre.treatment and 4-6 weeks after treatment
  Description: Depth of periodontal pockets measured at six sites per tooth using a PCPUNC-15 probe.
  Unit of Measure: Millimeters (mm)
Clinical Attachment Loss (CAL) | Pre-treatment and 4-6 weeks after treatment.
  Description: Distance from the cementoenamel junction to the base of the pocket.
  Unit of Measure: Millimeters (mm)
Periodontal Inflammation Severity Index (PIRIM, modified) | Pre-treatment and 4-6 weeks after treatment.
  Description: Calculated as the sum of periodontal pocket depth, normalized by the number of teeth.
  Unit of Measure: Index score (continuous variable, unitless)
Visible Plaque Index (VPI) | Pre-treatment and 4-6 weeks after treatment.
  Description: Proportion of sites with visible plaque. Unit of Measure: Percentage (%)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2025-02-01): https://cdn.clinicaltrials.gov/large-docs/84/NCT07200284/Prot_ICF_000.pdf